CLINICAL TRIAL: NCT03679585
Title: Talking Pictures: An Exploratory Study of a Meaning-Based Social Media Intervention for AYA Cancer Patients
Brief Title: Talking Pictures Social Media Intervention in Reducing Depressive Symptoms and Improving Spiritual Well-Being and Quality of Life in Adolescent and Young Adult Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: i 44717; NCI-2018-00023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 44717 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (social media intervention) (Experimental): Participants undergo Talking Pictures social media intervention for 10 weeks, receiving weekly assignments via email with requirements to use the Pixstori app to take and upload photographs with verbal narratives attached to a website. Participants can then share their pixstories to a group page and view and respond to others' pixstories.
  Interventions: Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Undergo Talking Pictures social media intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well Talking Pictures social media intervention works in reducing depressive symptoms and improving spiritual well-being and quality of life in adolescent and young adult cancer patients. Talking Pictures social media intervention may help doctors better learn how to most effectively provide psychosocial support to adolescent and young adult cancer patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and acceptability of a 10-week application (app)-based intervention.

II. To assess the impact of the intervention on depressive symptoms, spiritual well-being and quality of life.

III. To examine the content of participants recorded narratives for salient themes related to weekly content areas (e.g. identity, meaning-making, hopes, fears) in order to better understand the unique experiences and challenges of adolescent and young adult (AYA) patients.

OUTLINE:

Participants undergo Talking Pictures social media intervention for 10 weeks, receiving weekly assignments via email with requirements to use the Pixstori app to take and upload photographs with verbal narratives attached to a website. Participants can then share their pixstories to a group page and view and respond to others' pixstories.

After completion of study, participants are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and young adult cancer patients who were diagnosed within three years
* English comprehension in written and oral format
* Current possession of a smartphone, tablet, or computer with camera and wifi capacity or data plan
* Valid email address
* Pregnant women will be included if they meet eligibility requirements

Exclusion Criteria:

* Diagnosis of mental retardation, severe or untreated psychopathology (e.g. schizophrenia), or dementia
* Adults unable to consent: Will not include
* Prisoners will not be included given lack of access to smartphone

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Weekly photo task completion rate | At 10 weeks
  The observed completion rate will be described using the binomial completion proportion and its 2-sided 95% Jeffries confidence interval.
Project participation rates | At 10 weeks
  Study will be deemed feasible it least 11 of 30 participants demonstrate completion of assignments
Impact of intervention on depressive symptoms as assessed by Beck Depression Inventory-II (BDI-II) total score | Up to 2 months post intervention
  A series of repeated questionnaires will be conducted.
Impact of intervention on spiritual well-being as assessed by Functional Assessment of Chronic Illness Therapy Spiritual Well-Being (FACIT-Sp) total score | Up to 2 months post intervention
  A series of repeated questionnaires will be conducted.
Impact of intervention on psychosocial quality of life as assessed by Pediatric Quality of Life Inventory-Adolescent and Young Adult (PedsQL-AYA) psychosocial health score | Up to 2 months post intervention
  A series of questionnaires will be conducted.

SECONDARY OUTCOMES:
Participant satisfaction rating | At 10 weeks
  Satisfaction Questionnaire to be conducted

CONTACTS AND LOCATIONS:
Overall Officials: Megan Pailler, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States